CLINICAL TRIAL: NCT01939444
Title: A Pilot Study of the Bioavailability of Nasal Naloxone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OPI-12-001; 2012-004989-18 (EudraCT Number)
Record Dates: First submitted 2013-09-02; First posted 2013-09-11 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Drug Overdose
Keywords: Antidotes; naloxone; administration, intravenous; administration, intranasal; pharmacology
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- naloxone intranasal (Experimental): 2.0 mg by the nasal route
  Interventions: Drug: naloxone intranasal
- naloxone intravenous (Active Comparator): 1.0 mg intravenous
  Interventions: Drug: naloxone intravenous

INTERVENTIONS:
Drug: naloxone intranasal — If bioavailability is 20% or 50 %, the dose will be equivalent to the clinical range 0.4 - 1.0 mg given parenterally
  Arms: naloxone intranasal
Drug: naloxone intravenous — The parenteral dose reflects clinically used doses for overdoses (0.4 - 1.0 mg). A washout period of at least 3 days between each intervention. IV naloxone (Naloxone B. Braun 0.4mg/ml) administered slowly over 1-2 min in the recumbent position
  Arms: naloxone intravenous

SUMMARY:
The overall is aim of this pilot study is to give a preliminary estimation of key parameters of the pharmacokinetics of a proper formulation of intranasal naloxone. These data will be used to design a well justified protocol for the final estimation of these parameters:

* Preliminary estimation of bioavailability of this intranasal naloxone in human, healthy volunteers
* Preliminary estimation of the maximum serum concentration (Cmax) of this formulation
* Preliminary estimation of the time to maximum serum concentration (Tmax) of this formulation
* Safety of the formulation

ELIGIBILITY:
Inclusion Criteria:

* healthy (adequate organ function is determined by electrocardiogram (ECG), liver and kidney clinical chemistry, and a standard clinical examination/interview. For safety reasons we may ask for urine sample for analysis of opioids)
* informed consent

Exclusion Criteria:

* history of liver disease
* taking any medications including herbal medicines the last week history of drug abuse
* any local nasal disease or nasal surgery or recent cold for the last week
* any history of drug allergies

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
preliminary bioavailability of nasal naloxone | 2 weeks
  measured as ratio of area under the time concentration curve for nasal over intravenous naloxone x 100. Plasma concentration data will be analyzed by non-compartmental techniques.

SECONDARY OUTCOMES:
time to maximum concentrations | 2 weeks
maximum concentration | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ellingsen, MD PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of circulation and medical imaging, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Tylleskar I, Skulberg AK, Nilsen T, Skarra S, Dale O. Naloxone nasal spray - bioavailability and absorption pattern in a phase 1 study. Tidsskr Nor Laegeforen. 2019 Sep 23;139(13). doi: 10.4045/tidsskr.19.0162. Print 2019 Sep 24. English, Norwegian. PMID 31556537